CLINICAL TRIAL: NCT04029831
Title: Comparing the Effect of Different Ratio of Propofol-Ketamine Mixture (Ketofol) (6:1 vs. 4:1) for Sedation in Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: Comparison of Different Ratio of Ketofol (6:1 vs. 4:1) for Sedation in Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhrie Sugiarto, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes038
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K61 (Experimental): Patients in K61 group received propofol and ketamine in a ratio of 6:1. The 6:1 ketofol mixture was made by mixing 30 mL of 1% propofol (10 mg/mL) and 1 mL of ketamine (50 mg/ml), then 19 mL of 0.9% NaCl was added until the volume of the mixture was 50 mL. The 4:1 ketofol mixture was made by combining 20 mL of 1% propofol (10 mg/mL) and 1 mL ketamine (50 mg/ml). Afterward, 29 mL of 0.9% NaCl was added until the volume of mixture was 50 mL. Mixtures were mixed in a 50 mL syringe and were given to patients through a syringe pump (B Braun).
  Interventions: Drug: Propofol and Ketamine Mixture (Ketofol)
- K41 (Experimental): Patients in K41 group received propofol and ketamine in a ratio of 4:1. The 4:1 ketofol mixture was made by combining 20 mL of 1% propofol (10 mg/mL) and 1 mL ketamine (50 mg/ml). Afterward, 29 mL of 0.9% NaCl was added until the volume of mixture was 50 mL. Mixtures were mixed in a 50 mL syringe and were given to patients through a syringe pump (B Braun).
  Interventions: Drug: Propofol and Ketamine Mixture (Ketofol)

INTERVENTIONS:
Drug: Propofol and Ketamine Mixture (Ketofol) — Each group was given Ketofol, but group K61 received mixture of propofol and ketamine in a ratio of 6:1 while K41 received 4:1

SUMMARY:
Study was aimed to compare the effect of ketofol between 6:1 and 4:1 ratio in patients who underwent ERCP

DETAILED DESCRIPTION:
Combination of propofol and ketamine (ketofol) has been used as a medication for sedation in various medical procedures such as Endoscopic Retrograde Cholangio-pancreatography (ERCP). The addition of ketamine to propofol may counteract the effect of respiratory and cardiovascular depression of propofol. There has been limited studies evaluating the sedation effect of different ketofol dose ratios associated with hemodynamic changes, recovery time, dose and side effect. Thus, the study was aimed to compare the effect of ketofol between 6:1 and 4:1 ratio in patients who underwent ERCP

ELIGIBILITY:
Inclusion Criteria:

* Having ERCP procedures using sedatives
* ASA (American Society of Anesthesiologist) physical status Class I to III
* Body mass index (BMI) of 18-30 kg/m2
* Willing to participate in the study

Exclusion Criteria:

* Patients with a history of allergic reaction to medications used in the study
* Patients with cardiovascular disease, uncontrolled hypertension, respiratory dysfunction
* Patients with unstable hemodynamic
* Patients with psychiatric medications
* Patients with probability of difficult intubation and ventilation Patients with kidney disorder Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Level of Propofol Usage | 1 hour
  Level of propofol needed during the procedure

SECONDARY OUTCOMES:
Recovery Time | 15 minutes
  Time needed to recover after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coulter FL, Hannam JA, Anderson BJ. Ketofol dosing simulations for procedural sedation. Pediatr Emerg Care. 2014 Sep;30(9):621-30. doi: 10.1097/PEC.0000000000000222. PMID 25162687
- [Result] Bahrami Gorji F, Amri P, Shokri J, Alereza H, Bijani A. Sedative and Analgesic Effects of Propofol-Fentanyl Versus Propofol-Ketamine During Endoscopic Retrograde Cholangiopancreatography: A Double-Blind Randomized Clinical Trial. Anesth Pain Med. 2016 Aug 22;6(5):e39835. doi: 10.5812/aapm.39835. eCollection 2016 Oct. PMID 27853681